CLINICAL TRIAL: NCT02065271
Title: Herbal Preparation and Glucose Homeostasis
Acronym: Herbie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL44919.081.13
Record Dates: First submitted 2013-12-09; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Glucose Tolerance; Lipid Homeostasis; Vascular Function; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- herbal supplements (Experimental): 500mg, 3 per day, 4weeks
  Interventions: Dietary Supplement: herbal supplement
- placebo (Placebo Comparator): 500mg, 3 per day, 4 weeks
  Interventions: Other: placebo supplement

INTERVENTIONS:
Dietary Supplement: herbal supplement
  Arms: herbal supplements
Other: placebo supplement
  Arms: placebo

SUMMARY:
Rationale: The incidence of obesity and type 2 diabetes (T2D) is increasing rapidly and accounts for a considerable part of health care costs. Herbal supplements are used in many cultures for the prevention and treatment of many different conditions. Due to lack of scientific proof, the application in western cultures are minimal. Animal studies have shown that many constituents of such herbal supplements may have beneficial effects on several important parameters known to be affected in T2D. Still, no scientific proof in humans is available. We therefore aim to investigate the effect of 4-week herbal supplementation on glucose metabolism, lipid metabolism, vascular function and inflammation in subjects with increased fasting glucose levels or a decreased glucose tolerance.

Objective: The primary objectives are to investigate if 4-week herbal supplementation in subjects with increased fasting glucose levels or a decreased glucose tolerance has a positive effect on blood glucose levels and glucose tolerance. The secondary objectives are to investigate if 4-week herbal supplementation in subjects with increased fasting glucose levels or a decreased glucose tolerance has a positive effect on triglycerides (TG), total cholesterol (TC), low density lipoprotein (LDL), high density lipoprotein (HDL) levels, inflammation, adipose tissue and white blood cell gene-expression and AIX both fasted and during an OGTT test.

Study design: This study is a randomized, double-blind, placebo controlled cross-over trial in which two different treatments will be evaluated e.g. an intervention with the herbal mixture and a placebo. Each person will obtain both treatments in random order for four weeks with a wash out period of four weeks in-between. Fasting blood samples will be collected and subjects will receive a OGTT, paralleled by a PWA before and after 4-week supplementation.

Furthermore, after 4-week supplement intake we will collect a urine sample and collect an adipose tissue biopsy. The whole trial will last three months.

Study population: 26 overweight males and females 50-75yrs old with an increased fasting glucose or with an impaired glucose tolerance.

Intervention: Two intervention periods of 4-weeks in which participants will take three times a day a supplement of 500mg herbal or placebo.

Main study parameters/endpoints: Fasting blood glucose levels, glucose tolerance as determined by an oral glucose tolerance test (OGTT), AIX, triglycerides (TG), total cholesterol (TC), low density lipoprotein (LDL), high density lipoprotein (HDL) levels, PWA, adipose tissue an white blood cell gene expression and markers of inflammation .

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects that will participate in the study will invest a total of 16.5 hours. Blood collection by vena punctures/insertion of the venflon and the collection of an adipose tissue biopsy can occasionally cause a local hematoma or bruise and some participants may report pain or discomfort. The herbal supplements contain small amounts St. John's wort, which may affect the function of liver enzymes. We will therefore monitor liver function parameters during the supplementation period. Furthermore, subjects are excluded if they use medication known to be affected by St. John's wort. Participant will donate 284ml of blood, dispersed over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and postmenopausal females For females: menstrual cycle absent for more than 1 year
* age 50-70yrs
* BMI >27 kg/m2
* Increased fasting glucose or an impaired glucose tolerance (two-hour glucose levels >7.8 mmol/L on the 75-g oral glucose tolerance test or fasting glucose >6.1mmol/L).

Exclusion Criteria:

* Systolic blood pressure >160mmHg and diastolic blood pressure> 100mmHg
* Tobacco smoker
* Received inoculations within 2 months of starting the study or planned during the study
* Donated or intend to donate blood from 2 months before the study till months after the study.
* Unstable body weight (weight gain or loss >5kg in the past three months)
* Diagnosed with any long-term medical condition (e.g., diabetes, haemophilia, CVD, anemia, gastrointestinal disease, renal failure, thyroid disorders, cancer, HIV, hepatitis C)
* The use of the following medicine: medicine interfering with St Johns Worth such as, inhibitors of the immune system (ciclosporine, tacrolimus, everolimus, temsirolimus and sirolimus), coumarine type anticoagulant medicine (acenocoumarol and fenprocoumon), anti-epileptica (fenobarbital and fenytoïne), theophylline, atorvastatine, simvastatine, digoxine, kinidine, voriconazol, proton pump inhibitors (omeprazole and esomeprazole) and all anti-depressives ( incl. MAO inhibitors and SSRI's).
* Abuse of drugs/alcohol
* If the participant don't want to sign the informed consent
* If the participant don't want to be informed about unexpected findings during the screening or study
* Participation in another biomedical study
* Additional exclusion criteria for females:

Current use of contraceptives containing hormones Current use of hormone replacement therapy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change in glucose tolerance | baseline and after 4-week supplementation
  by oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
change in insulin | baseline and after 4-week supplementation
change in TAG | baseline and after 4 week supplementation
change in HbA1c | baseline and after 4 week supplementation
  glycosylated haemoglobin
change in FFA | baseline and after 4 week supplementation
change in cholesterol | baseline and after 4 week supplementation

OTHER OUTCOMES:
change in vascular function | baseline and after 4-week supplementation
  by pulse wave analysis (PWA)
change in ALAT/ASAT | baseline and after 4 week supplementation
Urinary metabolites | after 4 week supplementation
adipose tissue gene expression | after 4 week supplementation
  by qpcr
change in markers of inflammation | baseline and after 4 week of supplementation
  by PBMC genexpression and plasma cytokines

CONTACTS AND LOCATIONS:
Overall Officials: lydia a afman, phd, Study Director — Wageningen University
Locations (1):
- Wageningen university, Wageningen, Gelderland, Netherlands